CLINICAL TRIAL: NCT05596292
Title: Sensation of Dyspnea and Experience of Patients With Decompensated Heart Failure Undergoing an Early Mobilization Protocol With Immersive Virtual Reality: a Clinical Trial Protocol
Brief Title: Sensation of Dyspnea and Experience of Patients With Heart Failure
Acronym: MOVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-0355
Record Dates: First submitted 2022-10-07; First posted 2022-10-27 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Decompensated Heart Failure
Keywords: Early Mobilization; Cardiac Rehabilitation; Virtual reality; Exercise Tolerance; Patient experience

STUDY DESIGN:
Intervention Model Description: Single-center randomized parallel controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early mobilization protocol and immersive virtual reality (Experimental): Three days of an early mobilization protocol using immersive virtual reality glasses. The exercises will be progressed every day, starting in the first day with active movements of lower and upper limbs with cycle ergometer; in the second day repeat the first day exercise and do orthostasis training; and in the last day training ambulation. The immersive virtual reality glasses support a smartphone device, allowing videos to be used with 360º rotation and earpods headphones with bluetooth for sound. Video options will be offered to participants according to the exercise performed, ie: a cycling video for activities with a cycle ergometer; video with people walking for ambulation; and videos of the patient's choice, such as forest, beach or city scenarios, for other moments.
  Interventions: Device: Immersive Virtual Reality glasses; Other: early mobilization protocol
- early mobilization protocol (Active Comparator): Three days of an early mobilization protocol. The exercises will be progressed every day, starting in the first day with active movements of lower and upper limbs with cycle ergometer; in the second day repeat the first day exercise and do orthostasis training; and in the last day training ambulation.
  Interventions: Other: early mobilization protocol

INTERVENTIONS:
Device: Immersive Virtual Reality glasses — The immersive virtual reality glasses support a smartphone device, allowing videos to be used with 360º rotation and earpods headphones with bluetooth for sound. Video options will be offered to participants according to the exercise performed, ie: a cycling video for activities with a cycle ergometer; video with people walking for ambulation; and videos of the patient's choice, such as forest, beach or city scenarios, for other moments.
  Arms: early mobilization protocol and immersive virtual reality
Other: early mobilization protocol — Three days of an early mobilization protocol. The exercises will be progressed every day, starting in the first day with active movements of lower and upper limbs with cycle ergometer; in the second day repeat the first day exercise and do orthostasis training; and in the last day training ambulation.

SUMMARY:
This randomized clinical trial aims to evaluate patients with decompensated heart failure undergoing an early mobilization protocol with the use of immersive virtual reality glasses compared with patients undergoing the same protocol but without immersive virtual reality. The primary outcome will be the sensation of difficulty breathing, and the secondary outcome will be whether this technology provided a positive experience for patients in the intervention group that was superior to that of patients in the control group.

DETAILED DESCRIPTION:
This randomized clinical trial aims to assess the sensation of dyspnea in patients undergoing an early mobilization protocol with immersive virtual reality and their experience using this technology. The study population consists of patients with acute decompensated heart failure in an intensive care unit at a teaching hospital. The 3-day protocol will include active exercises with an in-bed cycle ergometer, orthostasis, and ambulation. The intervention group will perform all exercises using virtual reality glasses. The variables will be collected before and after each intervention.

ELIGIBILITY:
Inclusion Criteria - Patients with 18 years or older

* Being hospitalized for 24 hours or more
* Diagnosis of acute heart failure decompensated
* Being lucid and colaborative

Exclusion Criteria:

* Mechanical ventilation or circulatory support
* Neurodegenerative diseases
* Pregnant patients
* Hemodynamic instability at baseline
* Score on the Borg Rating of Perceived Exertion Scale Borg ≥ 4 at rest
* High risk of falls
* Difficulty communicating
* Not adapt with the immersive virtual reality glasses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline sensation of dyspnea on the Borg Rating Of Perceived Exertion Scale at immediately post-intervention | Up to 3 minutes before and up to 3 minutes after the early mobilization protocol with and without immersive virtual reality
  The evaluation of dyspnea sensation using the Borg Rating Of Perceived Exertion Scale. This scale has a score ranging from zero to 10, and the higher the score the patient reports, the greater the sensation of dyspnea

SECONDARY OUTCOMES:
Patient experience with and without immersive virtual reality during mobilization | Within 48 hours after the end of the early mobilization protocol with and without immersive virtual reality
  Assessment of patient experience using the Net Promoter Score, Likert and Analogical Scale

CONTACTS AND LOCATIONS:
Overall Officials: Eneida R Rabelo Silva, RN, MSc, ScD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Mobilization and experience data
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study Protocol when published
Access Criteria: When available

REFERENCES:
- [Derived] Caballero LG, Fraga IB, Tremea CEM, Perin G, Prates JDS, Lago PD, Oliveira JLC, Rabelo-Silva ER. Experience of heart failure patients in mobilization with virtual reality: mixed methods study. Rev Esc Enferm USP. 2025 Sep 15;59:e20250114. doi: 10.1590/1980-220X-REEUSP-2025-0114en. eCollection 2025. PMID 40955916
- [Derived] Fraga IB, Caballero LG, Lago PD, de Oliveira JLC, Scherer M, Haeffner MP, Rabelo-Silva ER. Perceived dyspnea and experience of hospitalized patients with acute decompensated heart failure undergoing an early MObilization protocol with immersive Virtual rEality: MOVE study protocol for a parallel superiority randomized clinical trial. Trials. 2023 Nov 24;24(1):751. doi: 10.1186/s13063-023-07786-z. PMID 38001540